CLINICAL TRIAL: NCT04850495
Title: A Phase Ib Trial of Zanubrutinib in Combination With R-PolaCHP (ZaR-PolaCHP) for Patients With Newly Diagnosed Diffuse Large B-Cell Lymphoma
Brief Title: Zanubrutinib in Combination With R-PolaCHP (ZaR-PolaCHP) for Newly Diagnosed Diffuse Large B-Cell Lymphoma
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Reached accrual limit
Sponsor: Yazeed Sawalha (Other)
Responsible Party: Sponsor-Investigator, Yazeed Sawalha, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20189; NCI-2021-01332 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Diffuse Large B-Cell Lymphoma; Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma; Transformed Marginal Zone Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Doxorubicin; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine; zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (zanubrutinib, R-CHOP) (Experimental): Patients receive zanubrutinib PO on days 1-21, rituximab IV on day 1, cyclophosphamide IV on day 1, doxorubicin hydrochloride IV on day 1, vincristine sulfate IV on day 1, and prednisone PO QD on days 1-5. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine Sulfate; Drug: Zanubrutinib

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
Drug: Zanubrutinib — Given PO
  Other Names: BGB-3111; Brukinsa; BTK-InhB

SUMMARY:
This phase Ib trial seeks to find out the best dose and possible side effects and/or benefits of zanubrutinib in combination with the R-PolaCHP in treating patients with newly diagnosed diffuse large B-cell lymphoma (DLBCL). Zanubrutinib is designed to block a protein called Bruton Tyrosine Kinase in order to stop cancer growth. R-CHOP is the acronym for the combination of five drugs: rituximab, cyclophosphamide, doxorubicin, vincristine and prednisone. It is the most widely used chemoimmunotherapy regimen for DLBCL and is considered the standard-of-care treatment for patients with DLBCL. Three of the drugs in R-CHOP (cyclophosphamide, doxorubicin and vincristine) are chemotherapy drugs. Rituximab is a type of immunotherapy and prednisone is a type of steroids.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the safety, toxicity profile and recommended phase 2 dose (RP2D) of zanubrutinib in combination with ZaR-PolaCHP (ZaR-PolaCHP) for patients with previously untreated diffuse large B-cell lymphoma (DLBCL).

SECONDARY OBJECTIVES:

I. Determine the objective response rate (ORR) (complete and partial responses), progression-free survival (PFS) and overall survival (OS) of ZaR-CHOP in patients treated at the RP2D.

II. Provide descriptive data on treatment exposure to zanubrutinib and R-CHOP including treatment discontinuation rate and relative dose intensity.

EXPLORATORY OBJECTIVES:

I. Examine archival tumor samples attained before starting treatment on trial to determine the clinical outcomes of molecularly defined DLBCL subtypes in patients treated with ZaR-Pola-CHP or ZaR-CHOP.

II. Measure circulating tumor deoxyribonucleic acid (DNA) (ctDNA) to correlate its presence with response by positron emission tomography (PET) imaging.

OUTLINE: This is a dose de-escalation study of zanubrutinib and fixed-dose R-CHOP regimen followed by a dose-expansion study.

Patients receive zanubrutinib orally (PO) once or twice daily on days 1-21, rituximab intravenously (IV) on day 1, cyclophosphamide IV on day 1, doxorubicin hydrochloride IV on day 1, vincristine sulfate IV on day 1, and prednisone PO QD on days 1-5. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed DLBCL, irrespective of cell-of-origin. Patients with previously diagnosed indolent lymphoma (follicular lymphoma and marginal zone lymphoma but not small lymphocytic lymphoma) who have transformed to DLBCL are eligible only if they have not previously been treated for indolent lymphoma except for local radiation for early-stage disease
* Patients may have received brief treatment with glucocorticoids (up to 250 mg/day prednisone or equivalent for a maximum of 10 days) and/or 1 cycle of chemotherapy such as R-CHOP (or some component[s] thereof) for the diagnosis of B-cell lymphoma provided they had staging computed tomography (CT) and/or positron emission tomography (PET)/CT scans prior to chemotherapy. Treatment must occur within 28 days prior to enrollment
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of zanubrutinib in combination with R-CHOP in patients <18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2. Performance status of 3 will be accepted if the impairment is caused by DLBCL complications and improvement is expected once therapy is initiated
* Measurable disease (defined as >= 1.5cm in diameter) or at least one PET fludeoxyglucose F-18 (FDG) avid area of disease
* Patients must have adequate hematologic, hepatic, and renal function as defined below:
* Hemoglobin >= 7.0 g/dL
* Absolute neutrophil count (ANC) > 1,000/mcL
* Platelet count > 75,000/mcL
* Total bilirubin =< 1.5 x the upper limit of the normal range (ULN) (unless due to Gilbert's disease)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) < 2.5 x institutional ULN
* Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) < 2.5 x institutional ULN
* Creatinine clearance > 40 mL/min calculated by Cockcroft-Gault
* Adequate cardiac function with a left ventricular ejection fraction (LVEF) >= 50% as assessed by echocardiogram or MUGA (Multigated acquisition scan)
* The effects of zanubrutinib on the developing human fetus are unknown. For this reason and because chemotherapeutic agents used in this study are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (double barrier method of birth control or abstinence) 2 weeks prior to initiation of treatment, for the duration of study participation and for 3 months after completing treatment. Should a woman become pregnant or suspect that she is pregnant while she or her partner is participating in this study, she should inform the treating physician immediately. Men must agree to refrain from sperm donation for at least 90 days after the last dose of zanubrutinib
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) or urine pregnancy test at screening. Women who are pregnant or breastfeeding are ineligible for this study
* Patients must have the ability to understand and the willingness to sign a written informed consent document and Health Insurance Portability and Accountability Act (HIPAA) consent document. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* International Prognostic Index must be documented:

  * ECOG performance status >= 2 (1 point)
  * Age >= 60 (1 point)
  * >= 2 extranodal sites (1 point)
  * Lactate dehydrogenase measurement (LDH) > upper limit of normal (1 point)
  * Ann Arbor Stage III or IV (1 point)
  * Is there evidence of transformation from indolent lymphoma?

Exclusion Criteria:

* Major surgery within 4 weeks before Day 1, Cycle 1 of treatment
* Prior anthracycline use >= 150 mg/m^2
* Known central nervous system (CNS) involvement. Patients at high risk for secondary CNS involvement but without neurologic symptoms suspected to be due to lymphoma are allowed to be enrolled and receive intrathecal chemotherapy with methotrexate, cytarabine, and/or glucocorticoids. Concurrent (during treatment with ZaR-polaCHP) CNS prophylaxis with IV methotrexate is NOT permitted in this study. CNS prophylaxis with IV methotrexate after completing ZaR-PolaCHP treatment and obtaining end-of-treatment response assessment is allowed. Patients who are enrolled and subsequently identified to have pathologic confirmation of CNS involvement by lymphoma may be continued on the study at the discretion of the principal investigator
* Active systemic bacterial, fungal or viral infection except for localized fungal infections of skin or nails. Patients with resolving infections such as urinary tract, respiratory, or skin infections may be enrolled if clinically improving. NOTE: patients may be receiving prophylactic antiviral or antibacterial therapies at the investigator's discretion
* Evidence of current uncontrolled or symptomatic cardiovascular conditions, including, uncontrolled cardiac arrhythmias, history of or symptomatic congestive heart failure (New York Heart Association [NYHA] Class III or greater), unstable angina, or myocardial infarction within the past 6 months. Poorly controlled or clinically significant atherosclerotic vascular disease including angioplasty, cardiac or vascular stenting within 6 months of enrollment
* History of cerebrovascular accident or transient ischemic attack within the 6 months before Day 1, Cycle 1 of treatment
* Any prior history of intracranial hemorrhage
* Known bleeding diatheses or platelet dysfunction disorders
* Known gastrointestinal (GI) disease or gastrointestinal procedure that will significantly interfere with the oral absorption or tolerance of zanubrutinib including the inability to swallow pills/capsules
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
* Evidence of prior malignancy except for: adequately treated non-melanoma skin cancer, adequately treated in situ carcinoma, low-grade prostate carcinoma (Gleason grade =< 6) managed with observation that has been stable for at least 6 months, or any malignancy treated with curative intent and continuously disease-free for at least 3 years
* Participation in other interventional clinical trials, including those with other investigational agents not included in this trial, within 21 days of Day 1, Cycle 1 of this trial. Also excluded are patients who are receiving any other investigational agents outside of a clinical trial
* Known history of human immunodeficiency virus (HIV), active hepatitis C infection (HCV ribonucleic acid [RNA] polymerase chain reaction [PCR]-positive) and/or active hepatitis B infections (HBV deoxyribonucleic acid [DNA] PCR-positive). If hepatitis B virus core (HBc) antibody is positive, the patient must be evaluated for the presence of HBV DNA by PCR. If HCV antibody is positive, the patient must be evaluated for the presence of HCV RNA by PCR. Patients with positive HBc antibody and negative HBV DNA by PCR are eligible. Patients with positive HCV antibody and negative HCV RNA by PCR are eligible
* Pregnant or breastfeeding women are excluded from this study. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with zanubrutinib, breastfeeding should be discontinued if the mother is treated with zanubrutinib. These potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 24 months
  Measured by the Common Terminology Criteria for Adverse Events version 5.0.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 5 years
  Defined as the proportion of patients achieving a complete or partial response. ORR will be reported with a 95% binomial confidence interval.
Progression-free survival | From the start of treatment to time of progression or death, whichever occurs first, assessed up to 5 years
  Will be estimated using the method of Kaplan-Meier, where the estimates at time points of interest will be reported with 95% confidence intervals.
Overall survival (OS) | From start of treatment to death from any cause, assessed up to 5 years
  Will be estimated using the method of Kaplan-Meier, where the estimates at time points of interest will be reported with 95% confidence intervals.
Zanubrutinib duration of treatment | Up to 6 cycles (each cycle is 21 days in length)
Zanubrutinib average daily dose | Up to 6 cycles (each cycle is 21 days in length)
Zanubrutinib discontinuation rate | Up to 6 cycles (each cycle is 21 days in length)
Zanubrutinib relative dose intensity | Up to 6 cycles (each cycle is 21 days in length)
  Defined as the ratio of the amount of a drug actually administered to the amount planned for a fixed time period.
Number of rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone (R-CHOP) cycles received | Up to 6 cycles (each cycle is 21 days in length)
R-CHOP discontinuation rates | Up to 6 cycles (each cycle is 21 days in length)
R-CHOP relative dose intensity | Up to 6 cycles (each cycle is 21 days in length)
  Defined as the ratio of the amount of a drug actually administered to the amount planned for a fixed time period.

CONTACTS AND LOCATIONS:
Overall Officials: Yazeed Sawalha, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - MUSC, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu